CLINICAL TRIAL: NCT02238496
Title: Pilot Trial of Temsirolimus and Perifosine in Recurrent/Progressive Malignant Gliomas
Brief Title: Perifosine and Torisel (Temsirolimus) for Recurrent/Progressive Malignant Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Andrew B Lassman, MD (Other)
Collaborators: Pfizer (Industry); AEterna Zentaris (Industry)
Responsible Party: Sponsor-Investigator, Andrew B Lassman, MD, John Harris Associate Professor of Neurology, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAM3801
Record Dates: First submitted 2014-08-29; First posted 2014-09-12 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Brain Tumor, Recurrent; Glioblastoma; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Mixed Glioma
Keywords: Glioblastoma; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Mixed Glioma; akt-Oncogene Protein; mTOR Protein; Glioma; Brain Neoplasms; Brain Tumor, Recurrent
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma | interventions — Cytoreduction Surgical Procedures; perifosine; temsirolimus

STUDY DESIGN:
Masking Description: No Masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Surgical Cohort - cytoreductive surgery (Other): Cytoreductive surgery planned (surgical cohort). After post-operative standard evaluations, patients will resume therapy. After anti-emetic prophylaxis, patients will receive the first divided dose of the perifosine loading dose after recovery from surgery. Patients will be observed for at least 30 minutes to ensure there has been adequate anti-emetic prophylaxis, and then patients will receive temsirolimus administered over 30-60 minutes IV. The remaining divided doses of the perifosine loading dose will then be administered. Patients will then return weekly for infusion of temsirolimus over 30-60 minutes IV. Dosing will be continuous although for the purposes of evaluation, a cycle will be defined as 4 weeks (28 days).
  Interventions: Procedure: Cytoreductive surgery; Drug: Perifosine; Drug: Temsirolimus
- Medical Cohort - no cytoreductive surgery (Other): No-Cytoreductive surgery planned (medical cohort). After anti-emetic prophylaxis, patients will receive the first divided dose of the perifosine loading dose. Patients will be observed for at least 30 minutes to ensure there has been adequate anti-emetic prophylaxis, and then patients will receive temsirolimus administered over 30-60 minutes IV. The remaining divided doses of the perifosine loading dose will then be administered. Patients will then return weekly for infusion of temsirolimus over 30-60 minutes IV. Dosing will be continuous although for the purposes of evaluation, a cycle will be defined as 4 weeks (28 days).
  Interventions: Drug: Perifosine; Drug: Temsirolimus

INTERVENTIONS:
Procedure: Cytoreductive surgery — Standard of care/routine cytoreductive glioma resection surgery. Arm B only.
  Other Names: Resection
  Arms: Surgical Cohort - cytoreductive surgery
Drug: Perifosine — Perifosine is a pill that has not been approved by the FDA which blocks a messenger that tells cancer cells to grow.
  Other Names: AEZS-104/D-21266; KRX-0401
Drug: Temsirolimus — Temsirolimus is an intravenous drug approved by the FDA for treatment of other cancers (kidney cancer, certain types of lymphoma) but not for brain tumors.
  Other Names: Torisel

SUMMARY:
The purpose of this study is to test the effectiveness of a drug called temsirolimus in combination with a drug called perifosine in treating brain tumors that have continued to grow after previous treatment. Temsirolimus is an intravenous drug approved by the FDA for treatment of other cancers (kidney cancer, certain types of lymphoma) but not for brain tumors. Perifosine is a pill that has not been approved by the FDA which blocks a messenger that tells cancer cells to grow. Research suggests that combined treatment with both drugs is better than either alone, and that it is reasonably safe.

DETAILED DESCRIPTION:
Malignant gliomas are the most common primary brain tumors, and glioblastoma (GBM) is the most common subtype in adults, representing more than 50% of gliomas. Standard initial treatment for newly diagnosed GBM consists of maximal surgical resection followed by radiotherapy to the tumor bed and chemotherapy with an oral DNA alkylator, temozolomide. However, recurrence is nearly universal despite standard therapy. There is no standard treatment at recurrence. Median survival is about 15 months from diagnosis and 6 months from recurrence. Once patients develop tumor progression, conventional chemotherapy is generally ineffective.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed intracranial glioblastoma (GBM), including sub variants
* At least 15 unstained slides or at least 1 tissue blocks must be collected from at least one prior surgery.
* Received prior radiotherapy and prior temozolomide as treatment for the malignant glioma
* Recovered from toxic effects of prior therapies and at least 2 weeks must have elapsed since any prior signaling pathway modulators; in general, at least 4 weeks must have elapsed from any other anticancer therapy
* Able to undergo contrast enhanced magnetic resonance imaging (MRI) scans or CT scans
* Shown unequivocal evidence for contrast enhancing tumor progression by MRI or CT in comparison to a prior scan
* Age > or = 18 years
* Karnofsky Performance Status > or = 70
* Life expectancy of > 8 weeks
* Normal organ and marrow function, adequate liver function, and adequate renal function before starting therapy
* Platelet count of at least 100,000/mm3 on at least 2 consecutive blood draws at least 1 week apart with results stable or trending upward
* Normal coagulation
* Cholesterol level < or = 350 mg/dl and triglycerides level < or = 400 mg/dl
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation
* Women of childbearing potential must have a negative beta-human chorionic gonadotropin (B-hCG) pregnancy test documented within 7 days prior to treatment
* Women must agree not to breast feed
* Ability to understand and the willingness to sign a written informed consent document
* Ability to swallow tablets

Group A (medical) specific inclusion criteria:

* Fulfill all of the general inclusion criteria
* At least 3 months between any prior brain radiotherapy and initiation of study therapy
* MRI/CT must demonstrate measurable enhancing tumor of at least 1cm squared in cross-sectional area to allow assessment of radiographic response
* On stable or decreasing dose of corticosteroids for a minimum of 5 days before the baseline MRI/CT
* The baseline brain MRI/CT must be performed less than 15 days prior to initiation of study treatment. Otherwise it must be repeated

Group B (surgical) specific inclusion criteria:

* Fulfill all of the general inclusion criteria
* Have cytoreductive surgery as part of their routine care for recurrent tumor
* Have cytoreductive surgery as part of their routine care for recurrent tumor
* A brain MRI/CT must be performed less than 15 days prior to initiation of study treatment. Otherwise it must be repeated

Exclusion Criteria:

* There is no limit on the number or type of prior chemotherapies except:

  1. convection enhanced delivery, catheter based intra-tumoral treatment, or carmustine (BCNU)/Gliadel® wafers
  2. stereotactic radiosurgery, or re-irradiation of any type
  3. agent designed to inhibit mTOR or PI3K/AKT
  4. direct Vascular Endothelial Growth Factor (VEGF)/Vascular Endothelial Growth Factor Receptors (VEGFR) inhibitors
* Smoking or plan to smoke tobacco or marijuana during study therapy
* Plan to eat grapefruit or drink grapefruit juice during study therapy
* Receiving any other investigational agents concurrently with study treatment
* Taking hepatic Enzyme Inducing Anti-Epileptic Drug (EIAED)
* Taking medications that are inducers or inhibitors of Cytochrome P450 3A4 (CYP3A4) for at least two weeks prior to study treatment
* Uncontrolled intercurrent illness
* HIV-positive patients on combination antiretroviral therapy
* Other active concurrent malignancy
* History of gout which can be exacerbated by perifosine
* Known history of allergic reactions attributed to compounds of similar chemical or biologic composition to temsirolimus or perifosine
* Therapeutic anticoagulation
* History of hemorrhagic or ischemic stroke
* Prior intratumoral bleeding must be evaluated with a non-contrast head CT to exclude acute blood prior to start of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2021-02-14 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit Rate | Up to 6 months from the start of treatment
  Clinical Benefit Rate is defined as the radiographic response rate plus 6-month progression-free survival (PFS) rate.

SECONDARY OUTCOMES:
Median Overall Survival Rate | Up to 48 months from start of treatment
  Overall survival will be calculated by using the interval between the date in which the first study drug administration took place (Arm A), and first day of study drug administration following surgery (Arm B), until the date of subject expiration.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B. Lassman, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Herbert Irving Comprehensive Cancer Center (HICCC) Clinical Trials Page — http://hiccc.columbia.edu/clinicaltrials